CLINICAL TRIAL: NCT04231448
Title: Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Tucidinostat in Combination With R-CHOP in Patients With Newly Diagnosed MYC/BCL2 Double-Expressor DLBCL
Brief Title: Phase III Study of Tucidinostat in Combination With R-CHOP in Patients With Newly Diagnosed Double-Expressor DLBCL
Acronym: DEB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDM302
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR-CHOP (Experimental)
  Interventions: Drug: R-CHOP(Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone); Drug: Tucidinostat
- R-CHOP (Placebo Comparator)
  Interventions: Drug: R-CHOP(Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone); Drug: Placebo

INTERVENTIONS:
Drug: R-CHOP(Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone) — R-CHOP : rituximab 375 mg/m2 IV, cyclophosphamide 750 mg/m2 IV, doxorubicin 50 mg/m2 IV, vincristine 1.4 mg/m2 IV [maximum total 2 mg], and prednisone [or equivalent] 100 mg orally as the background therapy for 6 cycles (21 days/cycle).
Drug: Tucidinostat — Tucidinostat ：30 mg was given orally after breakfast on day 1, day 4, day 8, day 11 in a 21-day cycle，for 6 cycles. After cycle 6 patients who are evaluated as complete response will receive 24 weeks additional administrations of Tucidinostat on day 1, day 4, day 8, day 11 in a 21-day cycle.
  Arms: CR-CHOP
Drug: Placebo — Placebo：30 mg was given orally after breakfast on day 1, day 4, day 8, day 11 in a 21-day cycle，for 6 cycles. After cycle 6 patients who are evaluated as complete response will receive 24 weeks additional administrations of placebo on day 1, day 4, day 8, day 11 in a 21-day cycle.
  Arms: R-CHOP

SUMMARY:
Tucidinostat (formerly known as chidamide) is an oral subtype-selective histone deacetylase inhibitor. This Randomized, Double-blind, Placebo-controlled Phase 3 trail is studying the efficacy and safety of Tucidinostat, in Combination with Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects With Newly Diagnosed MYC/BCL2 Double-Expressor Diffuse Large B-cell Lymphoma.

DETAILED DESCRIPTION:
The primary objective is to evaluate if the addition of Tucidinostat to rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) prolongs event-free survival (EFS) compared with R-CHOP alone in subjects with newly diagnosed MYC/BCL2 Double-Expressor subtype of DLBCL selected by IHC and FISH.

ELIGIBILITY:
Inclusion Criteria:

* Each potential subject must satisfy all of the following criteria to be enrolled in the study.

  1. Male or female, age ≥ 18 years and ≤80 years.
  2. No prior treatment for diffuse large B cell lymphoma(DLBCL), including hemotherapy, immunotherapy; radiotherapy (excluding local radiotherapy); monoclonal antibody therapy; surgical treatment (excluding biopsy)
  3. Histological or cytological confirmation of DLBCL

  <!-- -->

  1. CD20-positive DLBCL;
  2. Myc≥40% as well as Bcl-2≥50% through immunohistochemistry;
  3. Not with double (BCL-2 and c-MYC gene rearrangement) or triple (BCL-2, BCL-6, and c-MYC gene rearrangement) hit by FISH.

The verification of DLBCL will be based on local pathology report.15-20 unstained slides must be sent to the central laboratory for retrospective confirmation.

4.At least one positive lesion according to the Lugano Classification by fluorodeoxyglucose (FDG) positron emission tomography (PET)-computed tomography(CT).

5.Lymphoma International PrognosisIndex (IPI) score of 2,3,4. 6.Eastern Cooperative Oncology Group performance status grade of 0, 1, or 2. 7.Laboratory criteria are as follows except that caused by lymphoma assessed by the investigator (without receiving any supportive treatment for the following parameters within 2 weeks from the last dose prior to study entry):

(1)Hematology values:Hemoglobin (Hb)≥90g/L ; Absolute neutrophil count (ANC) ≥1.5×109/L ; platelets ≥90×109/L (2)Biochemical values: Serum creatinine ≤1.5×upper limit of normal(ULN); Total bilirubin ≤1.5 × ULN; Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) ≤2.5×ULN(ALT,AST≦5×ULN if liver involved).

8.Expected survival≥6 months. 9.All patients must have signed an informed consent document.

Exclusion Criteria:

* Any potential subject who meets any of the following criteria will be excluded from participating in the study.

  1. Presence of CNS involvement.
  2. Patients with primary DLBCL of the central nervous system (CNS),or secondary lymphoma of the central nervous system, or Primary mediastinal (thymic) large B-cell lymphoma, or Primary effusion lymphoma, or B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma, or Primary cutaneous DLBCL, leg type, or indolent lymphoma, or Burkitt lymphoma, or EBV-positive mucocutaneous ulcer, or DLBCL associated with chronic inflammation, or Lymphomatoid granulomatosis, or Intravascular large B-cell lymphoma, or ALK-positive large B-cell lymphoma, or Plasmablastic lymphoma, or HHV8-positive DLBCL, NOS, or primary testicular DLBCL.
  3. Patients with transformed lymphoma.
  4. History of organ transplantation or hematopoietic stem cell transplantation.
  5. Patients planned for autologous or allogeneic transplant as consolidation in first line.
  6. Patients with any other malignancy, except patients with a history of curatively treated basal or squamous cell carcinoma or in situ carcinoma of the cervix at any time prior to the study are eligible.
  7. Prior treatment with cytotoxic drugs for another condition (e.g., rheumatoid arthritis) or prior use of an anti-CD20 antibody within 5 years of the start of Cycle 1.
  8. Prior use of any monoclonal antibody within 3 months of the start of Cycle 1.
  9. Any investigational therapy within 3 months prior to the start of Cycle 1.
  10. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products.
  11. Contraindication to any of the individual components of CHOP.
  12. Corticosteroid use > 30 mg/day of prednisone or equivalent, for purposes other than lymphoma symptom control:

  <!-- -->

  1. Patients receiving corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to randomization (Cycle 1, Day 1).
  2. If glucocorticoid treatment is urgently required for lymphoma symptom control prior to the start of study treatment, prednisone 100 mg or equivalent could be given for a maximum of 5 days, but all tumor assessments must be completed prior to start of glucocorticoid treatment.

  13.Ongoing serious central nervous system disease or peripheral neuropathy, such as progressive multifocal leukoencephalopathy.

  14.Have uncontrolled or significant cardiovascular disease, including:
  1. Grade II or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (New York Heart Association Functional Classification ) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage.
  2. Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al).
  3. History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male), QTc≥470ms（female）at screening.
  4. Symptomatic coronary heart disease requiring treatment.
  5. Any other cardiovascular disease which is inappropriate for the study according to investigators' judgment.

  15.History of interstitial lung disease(ILD), or with ongoing signs and symptoms by CT or MRI at the time of screening.

  16.Patients with factors that could affect oral medication (such as dysphagia, chronic diarrhea, intestinal obstruction etc), or undergone gastrectomy.

  17.History of deep vein thrombosis or pulmonary embolism. 18.History of active bleeding within 2 months prior to the start of Cycle 1;or patients receiving anticoagulation therapy; or patients with evidence of bleeding potential according to investigators' judgment ( esophageal varices, active ulcer, or fecal occult blood test positive etc. ). Patients with bleeding led by lymphoma according to investigators' judgment are eligible.

19.6 weeks or less from the last major surgery that involved crucial organs, or with any other factors impede postoperative recovery according to investigators' judgment.

20.Known active infection, or active and uncontrolled hepatitis B infection(HBV), hepatitis C Virus(HCV), human immunodeficiency virus (HIV)/AIDS (Acquired Immune Deficiency Syndrome), or any other serious infection. (active infection defined as any major episode of infection requiring systemic treatment; Patients with occult or prior HBV may be included if HBV DNA is undetectable.) 21.Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or limit compliance with study requirements/ treatment.

22.Drug or alcohol abuse. 23.Women of childbearing potential and men who are sexually active not willing to practice a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials.These restrictions apply for 12 months after the last dose of rituximab or 12 weeks after the last dose of study drug, whichever is later. Pregnancy or lactation.

24.Any other condition which is inappropriate for the study according to investigators' judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | Up to approximately 5 years
  Defined as the duration from the date of randomization to the date of disease progression, relapse from CR , initiation of subsequent systemic antilymphoma therapy for residual disease, or death, whichever occurs first.

SECONDARY OUTCOMES:
Complete Response Rate(CRR) | Up to approximately 3 years
  Defined as the proportion of subjects with measurable disease who achieve CR.
Progression-Free Survival (PFS) | Up to approximately 5 years
  Defined as the duration from the date of randomization to the date of progression, relapse from CR, or death, whichever occurred first.
Overall Survival (OS) | Up to approximately 5 years
  defined as the duration from the date of randomization to the date of the participant's death
Disease-Free Survival (DFS) | Up to approximately 5 years
  Defined for patients achieving CR as the period from the date of the initial CR until the date of relapse or death from any cause.
Safety of Tucidinostat when combined with R-CHOP | Up to approximately 5 years
  All adverse events occurring during or after the first treatment will be summarized by treatment arm and NCI CTCAE grade.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Professor, Principal Investigator — Shanghai JiaoTong University School of Medicine，Ruijin Hospital; Jun Zhu, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai JiaoTong University School of Medicine，Ruijin Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No